CLINICAL TRIAL: NCT06698172
Title: Analysis of Motor Performance Improvement Following Visual Rehabilitation Treatment in Individuals with Visual Field Defects Due to Acquired Brain Injury
Brief Title: Motor Performance Improvement After Visual Rehabilitation
Acronym: VRvisual
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Carmen Lopez, Ph.D. from the University of Zaragoza, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRvisualfield
Record Dates: First submitted 2024-11-11; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Visual Field Loss; Balance; Brain Injury; Motor Performance
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VR Study Group (Experimental): Once the patient is included in the study, 12 weekly sessions of visual rehabilitation, each lasting 45 minutes, will be scheduled. A Virtual Reality device will be used along with the Visionary Sport visual therapy software.
  Interventions: Other: Virtual Reality rehabilitation

INTERVENTIONS:
Other: Virtual Reality rehabilitation — The study includes 12 weekly 45-minute visual rehabilitation sessions using a Virtual Reality device with Visionary Sport software. Originally designed for sports visual training, this software features gamified exercises to improve visual response times under professional supervision. Activities include games to enhance fixation, ocular motility, peripheral vision, and vergence.
  The "Peripheral Attention" activity trains reaction times to static stimuli perceived in the peripheral retina, adjustable to the patient's visual field defect. Stimuli can be placed at 10, 20, or 30 degrees in the peripheral field. The VR headset (Vive Focus 3) includes an eye tracker to monitor and adapt stimuli based on patient performance.
  Patients also perform 30 minutes of daily exercises at home, using proprietary software and Tobii 4C and 5C eye-tracking devices for ocular monitoring.

SUMMARY:
Acquired brain injury" refers to brain damage that impacts neurological processing, making daily activities challenging and often causing vision issues like binocular dysfunction, oculomotor problems, and visual field loss. In Spain, visual rehabilitation is limited, although it is more common in other countries.

These patients generally need an interdisciplinary approach involving professionals like physiotherapists and optometrists and often face mobility, balance, and spatial perception difficulties. Treatment tools include lenses, prisms, and technologies like virtual reality (VR). The Visionary VR program, presented by Dr. Portela, has shown promising results in visual field recovery by stimulating the affected area.

Visual rehabilitation is based on brain plasticity and involves three key strategies:

Prisms to expand the visual field. Compensatory therapy to improve eye movement. Restitution therapy to restore the visual field.

DETAILED DESCRIPTION:
Acquired brain injury is a term that covers all brain damage, and it is common for such an injury to have a profound effect on neurological processing. This can negatively impact how a person performs their daily activities. Many of these patients experience various vision problems alongside general health deterioration. A high percentage of individuals exhibit deficits in binocular fusion, oculomotor dysfunctions, and visual field loss (Ciuffreda, 2007). While visual rehabilitation for these patients is common in other countries, in Spain, these treatments within rehabilitation are usually only carried out occasionally.

Acquired brain injury can be due to various causes, including strokes, trauma, and tumours. It should be noted that due to the aging population, the number of strokes increases every year, and mortality from this cause is decreasing, leading to a growing number of patients with sequelae. Patients with brain injury may require rehabilitation treatment from various professionals, including physiotherapists, occupational therapists, speech therapists, and optometrists. Treatment in these cases should be interdisciplinary, considering the multiple disabling conditions these patients suffer from.

Since acquired brain injury can affect any area of the visual system, a rigorous evaluation of vision is necessary, paying attention to ocular health, visual function, motor function and binocular system, oculomotor skills, accommodative state, and the integrity of the visual field (Callahan, 2003).

In addition to visual field loss, patients with hemianopia may suffer from symptoms such as dizziness, vertigo, or nausea. There is also an increased risk of falls due to mobility issues, posture problems, gait variability, and balance, as well as difficulty navigating obstacles. Alterations in body schema and location can also occur, with this altered spatial perception impacting motor coordination, orientation, and object location (Kotecha, 2013).

Visual field loss can take different forms, including central loss, hemianopia, quadrantanopia, and altitudinal loss. Hemianopia refers to the loss of half the visual field, either right or left. Depending on the area of the visual pathway where the lesion occurs, bitemporal hemianopia, homonymous hemianopia, or superior/inferior quadrantanopia can develop. Quadrantanopia refers to the loss of a quadrant of the visual field. Visual field tests provide relevant information about the location of the brain lesion in these cases (Ruddy, 2022).

Furthermore, certain visual conditions are often overlooked, especially if they are mild, such as non-strabismic binocular vision dysfunctions, accommodative deficits, or ocular motility issues. If not considered, they can act as obstacles in the patient's rehabilitation, preventing them from performing various daily activities. Patients may sometimes suffer from diplopia, photophobia, or blurred vision, but in many cases, it is the difficulties they encounter in performing certain activities that indicate the presence of a visual problem. In patients with traumatic brain injury, it is estimated that 69% had at least one visual problem, mainly affecting accommodation, convergence, and ocular motility (Armstrong, 2018).

A stroke can cause some patients (20% to 57% of stroke patients) to lose the ability to see the entire space in front of them, often losing a whole half of the normal visual field. Ocular movement disorders can affect more than 70% of stroke patients, resulting in difficulties in maintaining both eyes in their normal position when looking straight ahead or in moving the eyes correctly to look in a different direction. This can affect the patient's depth perception, make it difficult to perceive the complete environment, and severely impact their reading ability.

These patients can benefit from visual treatment through compensatory lenses, compensatory prisms, visual field treatment, filters for photosensitivity, and visual rehabilitation aimed at improving the compromised visual skills. These treatments can be proposed in isolation or in combination during the patient's rehabilitation process (Armstrong, 2018; Thiagarajan, 2014; Thiagarajan, 2013; Gallaway, 2017).

Prisms are often used for fusional problems when the patient experiences diplopia or has difficulties performing convergence or divergence movements. They are also useful for visual field loss, projecting the image from the affected side of the visual field to the intact side. In this case, their goal is to expand or relocate the affected visual field, and they can be adapted binocularly or monocularly, either sectorially or across the entire lens.

Additionally, in the past year, Dr. Juan Portela, an optometrist, presented a novel treatment with a visual rehabilitation program using Virtual Reality at the II Neuro-Ophthalmology Conference in Valencia and the VII Low Vision Conference in October in Zaragoza. He achieved remarkable results in several patients with visual field loss using the Visionary virtual reality program (Visionary Sport, Gijón, Spain), increasing the visual field with stimuli appearing at the limit of the affected field area. This field restoration is reflected in visual field tests with fixation control in patients with hemianopia and altitudinal defects, which could have been caused by traumatic brain injury or stroke, even years before starting the Virtual Reality treatment. During the treatment, patient fixation was monitored using an eye tracker to control involuntary saccadic movements (Portela, 2023).

Previously, Casco et al. conducted a study using visual rehabilitation with Gabor patches in 10 patients with homonymous visual field defects for over six months, finding a significant improvement in the visual field, although it was approximately 5 degrees. The restored area improved letter recognition and the perception of moving shapes (Casco, 2018). Portela appears to have achieved better results in the cases he recently presented at several conferences.

Brain plasticity is the basis of visual rehabilitation, aiming to enhance the patient's visual skills and improve their quality of life as much as possible. The brain and its neural connections strengthen with the use of functions that depend on them. Visionary offers a set of exercises designed to rehabilitate deficits in visual tracking and binocular vision through perceptual learning. The Visionary software has been used in other studies related to visual rehabilitation in patients with amblyopia and limited stereopsis (Portela-Camino, 2018; Portela-Camino, 2021; Molina-Martín, 2020).

It is important to consider that there are three main strategies in the rehabilitation of patients with peripheral visual field loss, which can also be used in combination:

* Optical or substitution therapy using prisms. The goal is to expand the visual field by shifting part of the affected visual field to the healthy side of the field using the prism. Various strategies exist for this.
* Oculomotor or visual compensation therapy aims to enhance the patient's residual visual skills, improving the quality of ocular motility. This method helps the patient improve environmental scanning, first statically and then dynamically, with the ultimate goal of improving mobility. Visual-assisted therapy enhances outcomes for stroke patients with homonymous hemianopia alone or combined with oculomotor dysfunction. Visual therapy increased peripheral visual awareness. Additionally, patients felt safer in traffic and outdoor activities. Reading speed significantly increased, and the ability to keep a moving object in focus improved (Smaakjær, 2018).
* Visual field restitution therapy is based on cortical plasticity theories and the possibility of restoring the affected visual field (Casco, 2018).

The main objective of this project is to evaluate motor and balance improvement in patients with acquired brain injury and to analyse the improvement in the visual field following treatment with Virtual Reality.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects diagnosed with acquired brain injury either from a stroke or trauma.
* Subjects without cognitive impairment.
* Subjects without pre-existing musculoskeletal disorders prior to the acquired brain injury.
* Subjects without hemineglect.
* Subjects with more than 6 months of progression since the brain injury.
* Subjects who have an electronic device such as a computer and internet access to perform the exercises at home.
* Subjects with altitudinal visual field loss, hemianopia, or quadrantanopia with the central field preserved and at least 0.5 visual acuity.

Exclusion Criteria:

* Not signing the informed consent.
* Previous severe mental pathology to eliminate possible confounding factors if their daily activities are already affected.
* Uncontrolled epilepsy.
* Subjects with glaucoma or retinal pathologies affecting the visual field.
* Subjects with previous ocular surgery (cataract or refractive surgery) with less than 6 months of progression.
* Subjects who are not stable in any associated clinical pathology or otherwise diagnosed.
* Subjects who have previously undergone visual rehabilitation for the field defect.
* Not performing the proposed home exercises.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-29 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual field | 15 minutes
  The threshold test will be used in a 30-2 field size with fixation monitoring.
Balance | 15 minutes
  The stabilometric study will be conducted using the Podoprint® pressure platform (Grupo Namrol, Barcelona, Spain). A balance assessment will be conducted after 6 sessions and after 12 sessions of treatment.

SECONDARY OUTCOMES:
Visual Acuity | 2 minutes
  Measurement of visual acuity in near and distance vision
Subjective refraction | 5 minutes
  Evaluation of subjective refraction using trial lenses
Worth test | 1 minute
  The Worth Four Light Test is a clinical assessment of binocular vision, evaluating diplopia and suppression. The patient views a flashlight with four illuminated dots in a diamond pattern: one red at the top, two green on the sides, and one white at the bottom. The test is conducted at both 40 cm and 6 m distances.
Ramdom Dot 2 | 2 minutes
  This test is used to measure the patient's stereopsis between 900" and 12.5".
Cover Test | 1 minute
  The test requires the patient to focus on both a distant object and a near object at different times during the examination. An eye is covered briefly, then uncovered while observing any movement in both eyes. The cover test helps identify the type of ocular deviation and measures the degree of misalignment.
Maddox rod test | 1 minute
  The Maddox rod test is a subjective method for detecting and measuring latent or manifest strabismus by projecting a red line to one eye and a white light to the other, using prisms to determine the angle and amount of deviation.
Near point of convergence | 2 minutes
  The convergence test assesses a person's ability to focus on a near object, observing when diplopia (double vision) occurs and noting the point at which both eyes regain focus as the object is moved away.
Fusional vergences with prism bars | 4 minutes
  Fusional vergence was evaluated using a horizontal prism bar ranging from 1 to 40 prism diopters (pd) for both distance (6 m) and near fixations (40 cm). A single Snellen letter at the 6/12 level served as the fixation target for both distances. Prism strength was gradually increased, and patients indicated when the target appeared double. This prism strength was recorded as the break point, confirmed by the examiner as an exotropia without motor fusion recovery. The prism power was then reduced until the patient regained single vision, marking the recovery point. Both convergence and divergence break and recovery points were measured using base-out (BO) and base-in (BI) prisms, respectively.
Accommodative amplitude | 1 minutes
  The amplitude of accommodation will be measured using the push-up and push-down methods. It will be conducted in non-presbyopic patients.
Accommodative facility test | 3 minutes
  Monocular and binocular near accommodative facility will be measured using ±2.00 DS flipper at 40 cm. It will be conducted in non-presbyopic patients.
NSUCO test (Northeastern State University College of Optometry's Oculomotor test) | 2 minutes
  The NSUCO test assesses the quality of saccadic and pursuit eye movements. It provides a quick analysis with minimal patient cooperation. The setup involves two small colored reflective spheres (approximately 1/2 cm in diameter) on dowel sticks-one for pursuit and two for saccades.
DEM test (Developmental Eye Movement test ) | 3 minutes
  The DEM test evaluates the speed and accuracy of a participant's ability to read numbers in vertical and horizontal formats. It consists of a pretest and three test cards: two vertical subtests (A and B) with single-digit numbers, and one horizontal subtest (C) with more numbers in varying distances. The time taken for each subtest is recorded, and the ratio of horizontal to vertical time helps diagnose oculomotor dysfunction or difficulties in rapid automated naming.
DIVE device (Device for an Integral Visual Examination) | 3 minutes
  The DIVE device (Device for an Integral Visual Examination) is a digital tool developed to assess various aspects of visual function, particularly in children, including infants as young as six months and those with developmental challenges. It presents specialized visual stimuli on a high-resolution screen and uses eye-tracking technology to gather precise gaze data, allowing for automated and objective visual assessments.
Lawton and Brody Scale for Instrumental Activities of Daily Living (IADL) | 3 minutes
  The questionnaires will be applied to assess quality of life and daily activities before and after the intervention. Lawton and Brody Scale for Instrumental Activities of Daily Living (IADL) measures the degree of independence.
Barthel Index | 3 minutes
  The questionnaire will be applied to assess quality of life and daily activities before and after the intervention.
  • Barthel Index: Measures the ability of a person to perform ten daily activities, providing a quantitative estimate of their degree of independence. Scores range from 0 to 100, with lower scores indicating more dependence.
WHOQOL-BREF Questionnaire | 3 minutes
  The questionnaire will be applied to assess quality of life and daily activities before and after the intervention.
  • WHOQOL-BREF Questionnaire: A self-administered instrument that provides a profile of perceived quality of life, consisting of 26 questions developed from the original 100-section version (Whoqol-100).

CONTACTS AND LOCATIONS:
Overall Officials: Maria José López de la Fuente, PhD, Study Chair — Universidad de Zaragoza; Jorge Pérez Rey, PhD, Study Chair — Universidad de Zaragoza; Naiara Díaz Marín, MSc, Study Chair — Universidad de Zaragoza; Javier Mateo Gabás, PhD, Study Chair — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No